CLINICAL TRIAL: NCT07012785
Title: Efficacy Analysis of Saccharomyces Boulardii Combined With Minocycline in Treatment-naïve Patients With Helicobacter Pylori Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Chen Lu, Director, Zhongda Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025ZDSYLL071-P01
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Drug: Bismuth quadruple therapy
- Experimental group (Experimental)
  Interventions: Drug: Saccharomyces boulardii

INTERVENTIONS:
Drug: Bismuth quadruple therapy — Bismuth quadruple therapy
  Arms: Control Group
Drug: Saccharomyces boulardii — Saccharomyces boulardii
  Arms: Experimental group

SUMMARY:
To assess the efficacy and safety of Saccharomyces boulardii combined with triple therapy containing minocycline in the initial eradication of Helicobacter pylori (H. pylori) infection

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years, regardless of gender;
2. Positive 13C/14C urea breath test result;
3. No previous history of H. pylori eradication treatment;
4. Agreement to participate in this study and signing of the informed consent form.

Exclusion Criteria:

1. History of ≥ 1 instance of failed H. pylori eradication;
2. Use of antibiotics (including antibacterial traditional Chinese medicines), nonsteroidal anti-inflammatory drugs (NSAIDS), bismuth agents, H2 receptor antagonists (H2RAs), proton-pump inhibitors (PPIs), and potassium-competitive acid blockers (P-CAB) within 4 weeks before treatment;
3. Plans to conceive, pregnancy, or breastfeeding;
4. Severe liver, kidney, or cardiovascular diseases; malignancies; and alcoholism;
5. Allergies to the drugs used in this study or a history of penicillin allergy;
6. The inability to correctly express one's symptoms and wishes, such as inability due to mental illness or severe neurosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
H. Pylori eradication rate | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China